CLINICAL TRIAL: NCT03933982
Title: Pyrotinib Plus Vinorelbine in Patients With Brain Metastases From HER2-positive Metastatic Breast Cancer : a Prospective, Single-arm, Open-label Study
Brief Title: A Study of Pyrotinib Plus Vinorelbine in Patients With Brain Metastases From HER2-positive Metastatic Breast Cancer
Acronym: Pyrotinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC1865
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer; Brain Metastases
Keywords: Breast cancer, Brain metastases, Pyrotinib, Vinorelbine, HER2
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — pyrotinib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib plus Vinorelbine (Experimental)
  Interventions: Drug: Pyrotinib Plus Vinorelbine

INTERVENTIONS:
Drug: Pyrotinib Plus Vinorelbine — Pyrotinib: 320mg/d, q.d., p.o. A course of treatment need 21 days. Vinorelbine: 60mg/m2 q.d. d1,8,15, p.o. A course of treatment need 21 day.

SUMMARY:
Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER1, HER2 and HER4 receptors. This study is a single-arm, prospective, open label clinical study of pyrotinib plus vinorelbine as the therapy of brain metastases from HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age18-75 years.
2. ECOG performance status ≤2.
3. Histologically confirmed HER2 positive advanced breast cancer.
4. Prior to anthracyclines and taxanes (neoadjuvant, adjuvant and metastatic setting). Received ≤4 regimes in metastatic setting. Prior to trastuzumab is allowed.
5. Not received whole brain radiotherapy (WBRT) or recurrence after WBRT.
6. Controlled CNS symptoms (headache, dizziness, lethargy, nausea etc.).
7. Patients with CNS metastasis; at least one CNS metastases with a longest diameter ≥1 cm and a diameter perpendicular to the longest diameter should be ≥0.5 cm;
8. Signed the informed consent form prior to patient entry.

Exclusion Criteria:

1. Participated in other drug clinical trials within 4 weeks before the start of the study;
2. Received radiotherapy, chemotherapy, surgery and target therapy within 4 weeks before the start of the study;
3. Received endocrine therapy within 7 days before the start of the study;
4. Suitable for surgical resection;
5. Accompanied by rapid progress of organ invasion;
6. Factors influencing the usage of oral administration (such as unable to swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction etc.).
7. Prior to pyrotinib or vinorelbine or anti-HER2 TKI drugs;
8. Allergies to any compounds of experimental drugs;
9. CNS disorders or mental disorders, history of clear neurological or mental disorders, including epilepsy or dementia;
10. Other malignancies within 5 years, except cured in-situ of uterine cervix carcinoma , skin basal cell carcinoma and squamous-cell carcinoma.
11. Any other situations judged by investigator as not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-22 (Actual); Primary Completion 2021-12-22 (Estimated); Study Completion 2022-06-22 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) of CNS | Estimated up to 1 year
  ORR, defined as proportion of complete response and partial response according to RANO-Brain Metastases (RANO-BM) criteria.

SECONDARY OUTCOMES:
Time to progression (TTP) | Estimated up to 1 year
  TTP, defined as the time from the date of informed consent until the date of disease progression (PD), either CNS PD or extracranial PD, whichever comes first.
OS (overall survival) | Estimated up to 1 year
  OS, defined as the time from the date of informed consent until to the date of death, regardless of the cause of death.
Time to radiotherapy | Estimated up to 1 year
  Time to radiotherapy, defined as the time from the date of informed consent until to the date of radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, M.D., Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No